CLINICAL TRIAL: NCT07329751
Title: Based on the Spatio-temporal Coding Characteristics of Frontotemporal Network, This Paper Explores the Mechanism of Five-tone Speech Training in Reshaping Language Fluency Function.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ruiming Nan, Professor, Fujian University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jia Huang
Record Dates: First submitted 2025-09-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Aphasia
Keywords: aphasia; stroke; pentatonic scales of chinese medicine
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group for Traditional Chinese Medicine Pentatonic Sound Therapy (Experimental): Therapeutic Protocol for 'Five-Tone' Therapy Based on Melodic Intonation Training Model: Subjects undergo syndrome differentiation and treatment, with corresponding 'Five-Tone' melodies selected for active training based on the melodic intonation intervention model. Intervention duration: All eligible participants in this study received four weeks of treatment, administered once daily for 40 minutes, five days per week.
  Interventions: Other: Traditional Chinese Medicine Five-Tone Therapy
- Melodic Intonation Therapy Treatment Group (Active Comparator): Melodic intonation training. Intervention duration: All eligible participants enrolled in this study received treatment for 4 weeks, once daily for 40 minutes, with sessions conducted 5 days per week.
  Interventions: Other: Melodic Intonation Training
- Conventional control group (Active Comparator): ① Rehabilitation training: Physicians conduct limb movement and speech rehabilitation training for participants in accordance with the Clinical Evidence-Based Practice Guidelines for Integrated Traditional and Western Medicine Rehabilitation of Stroke (2024 Edition). ② Conventional Medical Management: Standard foundational treatment is administered to enrolled subjects in accordance with the National Health Commission's Guidelines for the Prevention and Treatment of Cerebrovascular Diseases (2024 Edition). This encompasses: management of underlying causes, blood pressure control, antiplatelet therapy, anticoagulant therapy, and regulation of blood glucose and lipid levels. ③ Health Education: Health education is provided to subjects to raise awareness of the severe risks associated with stroke and the available rehabilitation interventions.
  Interventions: Other: Standard speech therapy; Routine medical treatment; Health education

INTERVENTIONS:
Other: Traditional Chinese Medicine Five-Tone Therapy — Therapeutic Protocol for 'Five-Tone' Therapy Based on Melodic Intonation Training Model: Subjects undergo syndrome differentiation and treatment, with corresponding 'Five-Tone' melodies selected. Based on the melodic intonation training model, active training is conducted through melodic intervention measures. ① Rehabilitation training② Conventional Medical Management.③ Health Education:
  Arms: Experimental Group for Traditional Chinese Medicine Pentatonic Sound Therapy
Other: Melodic Intonation Training — All eligible participants enrolled in the study received four weeks of melodic intonation therapy, administered once daily for 40 minutes, five days per week.① Rehabilitation training② Conventional Medical Management.③ Health Education:
  Arms: Melodic Intonation Therapy Treatment Group
Other: Standard speech therapy; Routine medical treatment; Health education — ① Rehabilitation training: Physicians conduct limb movement and speech rehabilitation training for participants in accordance with the Clinical Evidence-Based Practice Guidelines for Integrated Traditional and Western Medicine Rehabilitation of Stroke (2024 Edition). ② Conventional Medical Management: Standard foundational treatment is administered to enrolled subjects in accordance with the National Health Commission's Guidelines for the Prevention and Treatment of Cerebrovascular Diseases (2024 Edition). This encompasses: management of underlying causes, blood pressure control, antiplatelet therapy, anticoagulant therapy, and regulation of blood glucose and lipid levels. ③ Health Education: Health education is provided to subjects to raise awareness of the severe risks associated with stroke and the available rehabilitation interventions.
  Arms: Conventional control group

SUMMARY:
To explore the mechanism of five-tone speech training in reshaping language fluency function and the clinical efficacy of aphasia language function, daily communication ability and communication efficiency based on the temporal and spatial coding characteristics of frontotemporal network. Combined with EEG ( rsEEG, ERP ), nuclear magnetic resonance examination and near-infrared imaging system examination to explore its effect on brain electrophysiological activity. So as to promote the modernization of traditional Chinese medicine rehabilitation treatment technology and the popularization and application of speech rehabilitation treatment technology.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Age between 18 and 70 years

Right-handed

Native Chinese speakers

Clinical diagnosis of post-stroke aphasia caused by ischemic stroke, confirmed by CT or MRI

Diagnosis of non-fluent aphasia based on the Western Aphasia Battery (WAB), with BDAE severity rating of 1-5

Time since stroke onset ≥ 2 weeks

Stable vital signs, clear consciousness, and no severe cognitive impairment

Ability to understand the study procedures and provide written informed consent (or consent provided by a legally authorized representative)

Exclusion Criteria:

History of aphasia or neurological disease not caused by stroke (e.g., traumatic brain injury, brain tumor, neurodegenerative diseases)

Severe visual or auditory impairments that would interfere with task performance

Severe cognitive impairment or disorders of consciousness preventing cooperation with language assessment or intervention

Severe dysarthria or apraxia of speech that precludes valid language assessment

History of epilepsy or other severe neurological conditions

Severe systemic diseases (e.g., severe cardiopulmonary dysfunction, renal failure, hepatic failure, malignancy)

Psychiatric disorders (e.g., schizophrenia, severe depression, or other major psychiatric illnesses)

Contraindications to MRI or fNIRS assessment (e.g., metallic implants, severe claustrophobia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Semantic Fluency Test | Baseline and Week 4 post-intervention
  The semantic fluency test requires subjects to say as many words related to a given semantic category as possible within 60 seconds, such as furniture, occupation, etc. The more words they say, the better the surface semantic fluency.
Speech fluency test | Baseline and Week 4 post-intervention
  Verbal Fluency Test: Participants are required to produce as many words as possible within 60 seconds that belong to a specified phonetic category, such as words beginning with "yi". A higher number of words indicates greater apparent verbal fluency

SECONDARY OUTCOMES:
Boston Diagnostic Aphasia Examination，BDAE | Baseline and Week 4 post-intervention
  BDAE Aphasia Severity Grading Scale ranges from 0 to 5, with higher grades indicating better language ability.
  Grading and Language Performance Grade 0: No meaningful speech; no auditory comprehension. Grade 1: Discontinuous speech in communication, but mostly requiring listeners to infer, ask questions, and guess; limited scope of communicable information; listeners find verbal communication difficult.
  Level 2: With listener assistance, conversation on familiar topics may be possible. However, expressing thoughts on unfamiliar subjects is often impossible, causing difficulty for both patient and examiner.
  Level 3: With minimal or no assistance, the patient can discuss nearly all everyday matters. Yet, due to diminished verbal and/or comprehension abilities, certain conversations prove difficult or unlikely.
  Level 4: Speech is fluent, though perceptible comprehension difficulties may be noted. Thought and verbal expression remain largely unrestricted.
  Level 5: Minimal discernible spee
Minimum Mental State Examination | Baseline and Week 4 post-intervention
  MMSE total score: 30 points
  1. Cognitive impairment: Maximum score 30 points; scores 27-30 indicate normal cognition, while scores <27 indicate cognitive impairment.
  2. Dementia classification criteria:
     Illiterate ≤ 17 points Primary education ≤ 20 points Secondary education (including technical secondary) ≤ 22 points Tertiary education (including college) ≤ 23 points
  3. Dementia severity grading:
  Mild: MMSE ≥ 21 points Moderate: MMSE 10-20 points Severe: MMSE ≤ 9 points The Mini-Mental State Examination assesses cognitive function. The scale ranges from 0 to 30 points, with higher scores indicating better cognitive function.
Western Aphasia Battery，WAB | Baseline and Week 4 post-intervention
  The Western Aphasia Battery Aphasia Quotient (AQ) is calculated from four component scores: spontaneous speech, auditory comprehension, repetition, and naming, with a maximum total of 100 points. An AQ score below 93.8 indicates diagnostic aphasia. The assessment comprises four major components: spontaneous speech (20 points total, divided into information content 10 points and flow 10 points), listening comprehension (10 points), repetition (10 points), and naming (10 points). The Aphasia Quotient (AQ) is then calculated. A higher Aphasia Quotient indicates better language ability.
Chinese Functional Communication Profile, CFCP | Baseline and Week 4 post-intervention
  Scale Name: Functional Language Communication Ability Assessment Scale Score Range: 0 to 100 points Score Interpretation: Higher scores indicate better functional communication abiity.
  'The Functional Language Communication Ability Assessment Scale evaluates patients' practical communication skills in everyday life situations. The scale's total score ranges from 0 to 100 points, with higher scores representing superior functional communication ability.'

IPD SHARING:
Plan to Share IPD: No
Data sharing will be subject to strict limitations to comply with the General Data Protection Regulation (GDPR), HIPAA (where applicable in the United States), and other relevant data privacy regulations. Neither our agreement with the Ethics Committee nor the participants' informed consent forms envisage data being shared broadly for purposes beyond the specific analysis plan of this trial.